CLINICAL TRIAL: NCT06901388
Title: Peri-implant Disease Perception Before and After Non-Surgical Peri-implant Therapy: A Pre-post Quasi-Experimental Study
Brief Title: Peri-implant Disease Perception Before and After Non-Surgical Peri-implant Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Nicola Discepoli, Associate Professor, University of Siena
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BIPP001
Record Dates: First submitted 2025-03-22; First posted 2025-03-28 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Peri-implant Mucositis; Peri-Implantitis
Keywords: Oral Health Impact Profile 14; Brief-Illness Perception Questionnaire; Non-surgical peri-implant therapy
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group (Experimental): All participants will receive non-surgical peri-implant therapy consisting of mechanical debridement and oral hygiene instruction. Psychometric assessments (Brief-IPQ and OHIP-14) will be administered at baseline and 3 months after treatment to evaluate changes in illness perception and oral health-related quality of life.
  Interventions: Procedure: Non-surgical peri-implant therapy

INTERVENTIONS:
Procedure: Non-surgical peri-implant therapy — Standardized non-surgical therapy consisting of mechanical debridement of peri-implant sites using ultrasonic instruments, combined with personalized oral hygiene instruction. The intervention is delivered in a single session. No adjunctive antimicrobials are used. Follow-up is scheduled 3 months after therapy for clinical and psychometric re-evaluation.
  Other Names: Mechanical debridement + Oral hygiene instruction

SUMMARY:
The present pre-post quasi-experimental study assessed changes in peri-implant disease perception and oral health-related quality of life following non-surgical peri-implant therapy. Using validated psychometric tools, including the Brief Illness Perception Questionnaire (Brief-IPQ) and the Oral Health Impact Profile-14 (OHIP-14), the study evaluates patients at baseline and three months after therapy. The study builds upon prior cross-sectional findings highlighting the low perception of peri-implant diseases and aims to determine whether non-surgical treatment improves patients' psychological awareness and perceived impact of their condition.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 80 years
* Diagnosis of peri-implant disease requiring non-surgical therapy
* Presence of at least one dental implant loaded for a minimum of one year
* History of periodontitis
* Good general health
* Ability to provide written informed consen

Exclusion Criteria:

* Pregnant or lactating individuals
* Inability to perform basic oral hygiene procedures
* Inability to understand or complete study questionnaires

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2025-03-31 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
Change in illness perception (Brief-IPQ total score) | Baseline and 3 months from baseline
  Illness perception will be assessed using the Brief Illness Perception Questionnaire (Brief-IPQ). The primary outcome is the change in the total score from baseline to 3 months after baseline, following non-surgical peri-implant therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- AOUS, Siena, Italy